CLINICAL TRIAL: NCT02533271
Title: Phase III Study of Short-term Radiotherapy Plus Neoadjuvant Chemotherapy Versus Preoperative Long-term Chemoradiotherapy in Locally Advanced Rectal Cancer
Brief Title: Optimization of Preoperative Treatment in Locally Advanced Rectal Cancer
Acronym: STELLAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., vice director of Radiotherapy Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XT2015-03; CH-GI-090 (Other: Ethics Committee of Cancer Institute and Hospital, Chinese Academy of Medical Sciences)
Record Dates: First submitted 2015-08-21; First posted 2015-08-26 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cancer, Rectum
Keywords: rectal cancer; short-term radiotherapy; neoadjuvant chemotherapy; total mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNT group (Experimental): The intervention of TNT group is Short-course radiotherapy with neoadjuvant chemotherapy, which consists of a short-course radiotherapy (SCRT, 5 Gy x 5 alone), then after 7-10 days of radiotherapy completed, patients will receive neoadjuvant chemotherapy, given in 3 week cycle of capecitabine 1000 mg/m2 twice daily, day 1-14 combined with oxaliplatin 130 mg/m2 once. In total, 4 cycles of neoadjuvant chemotherapy are prescribed preoperatively, then followed by a total mesorectal excision(TME) and postoperative adjuvant chemotherapy. If patients are eligible for postoperative chemotherapy this should consist of at least 2 cycles, which are the same as neoadjuvant chemotherapy.
  Interventions: Radiation: Short-course radiotherapy with neoadjuvant chemotherapy
- CRT group (Other): The intervention of CRT group is long-term chemoradiotherapy(CRT), which consists of a long-term chemoradiation (2 Gy x 25 with capecitabine) preoperatively, followed by a total mesorectal excision(TME) and then postoperative adjuvant chemotherapy. The radiotherapy is given in combination with capecitabine in a dose of 825 mg/m2 twice daily on days when radiotherapy, excluding weekends. If patients are eligible for postoperative chemotherapy this should consist of at least 6 cycles of capecitabine 1000 mg/m2 twice daily, day 1-14 combined with oxaliplatin 130 mg/m2 once every 3 weeks.
  Interventions: Radiation: Long-term chemoradiotherapy

INTERVENTIONS:
Radiation: Short-course radiotherapy with neoadjuvant chemotherapy — Short-course radiotherapy with 4 cycles of neoadjuvant chemotherapy
  Arms: TNT group
Radiation: Long-term chemoradiotherapy — Standard chemoradiotherapy
  Arms: CRT group

SUMMARY:
The purpose of this study is to compare effectiveness of short-term radiotherapy with neoadjuvant chemotherapy(TNT group) with preoperative long-term chemoradiotherapy(CRT group) in locally advanced rectal cancer. The hypothesis is 3-year disease-free survival in TNT group was non-inferior to that in CRT group.

DETAILED DESCRIPTION:
The study is a prospective phase III randomized multicenter trial. The purpose of this study is to compare short-term radiotherapy with neoadjuvant chemotherapy(TNT group) with preoperative long-term chemoradiotherapy(CRT group) for middle-lower locally advanced rectal cancer. The primary endpoint is 3-year disease-free survival,defined as the interval from randomization to the first occurrence of local-regional failure, distant metastasis, second primary tumor or death from any cause. The primary hypothesis was that DFS in the TNT group would be non-inferior to that in the CRT group. After preoperative radiotherapy and surgery, the DFS rate of LARC fluctuated from 50% to 65%. Assuming a 3-year DFS rate in CRT group is 65%, we consider the 3-year DFS rate in the TNT group is not lower than 54% (e.g., a margin of 11% or equivalently, hazard ratio (HR) < 1.43). Guarding against a 5% ineligibility or drop-out rate, the accrual target was 600 patients, with the final analysis to occur after at least 194 DFS events to provide at least 80% power at 1-sided type 1 error of 0.05. The choices of type 1 error and power were made to provide an appropriate comprise between feasibility, timeliness and statistical rigor of evidence generation.

This study seeks to compare outcomes between two groups with respect to rates of overall survival(OS), distance metastasis free survival (DMFS), and locoregional recurrence free survival (LRRFS).In addition, acute and late toxicity profile, completion of preoperative treatment, the proportion of patients with radical resection (R0), surgical complication profile, the rate of pathological complete response (pCR), and quality of life (QoL) are also secondary endpoints.

The STELLAR-trial has been designed by National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, and the hypothesis is 3-year disease-free survival in TNT group was non-inferior to that in CRT group.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven rectal adenocarcinoma;
* Distance between tumour and anal verge≤ 10cm;
* Locally advanced tumour;(AJCC Cancer Staging:T3, T4 or N+)
* Cancer Staging must be based on pelvic MRI;
* Eastern Cooperative Oncology Group(ECOG) performance score ≤ 1;
* Written informed consent;
* Mentally and physically fit for chemotherapy;
* Adequate blood counts: White blood cell count ≥3.5 x 109/L Haemoglobin levels ≥100g/L Platelet count ≥100 x 109/L Creatinine levels ≤1.0× upper normal limit（UNL） Urea nitrogen levels ≤1.0× upper normal limit（UNL） Alanine aminotransferase(ALT) ≤1.5× upper normal limit（UNL） Aspartate aminotransferase(AST) ≤1.5× upper normal limit（UNL） Alkaline phosphatase(ALP) ≤1.5× upper normal limit（UNL） Total bilirubin(TBIL) ≤1.5× upper normal limit（UNL）
* No excision of tumor, chemotherapy or other anti-tumor treatment after the diagnosis.

Exclusion Criteria:

* Distant metastases;
* Recurrent rectal cancer;
* Active Crohn's disease or ulcerative colitis;
* Concomitant malignancies;(except basocellular carcinoma or in-situ cervical carcinoma)
* Allergic to Fluorouracil or Platinum drugs;
* Contraindications to MRI for any reason;
* Concurrent uncontrolled medical condition;
* Pregnancy or breast feeding;
* Known malabsorption syndromes or lack of physical integrity of upper gastrointestinal tract;
* Symptoms or history of peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-08; Primary Completion 2023-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | three year

SECONDARY OUTCOMES:
Overall survival rate | three year
Distance metastasis free survival rate | three year
Locoregional recurrence free survival rate | three year
Incidence of surgical complications | one month
  Surgical complications are defined as those occurring within 30 days after surgery, such as re-operation, anastomotic fistula, bleeding, infection and death related to the operation, etc.
Incidence of acute toxicities during radiation or chemotherapy | three months
  Number of participants with abnormal laboratory values and/or adverse events that are related to radiation or chemotherapy as assessed by Common Toxicity Criteria for Adverse Effects(CTCAE) v4.0.
Radical resection (R0) | one year
  R0 resection rate is R0 resection probability of radical surgery in patients with locally advanced rectal cancer after neoadjuvant therapy
The rate of pathological complete response (pCR) | one year
  PCR rate is pathological ypT0N0 probability of radical surgery in patients with locally advanced rectal cancer after neoadjuvant therapy
Quality of life (QoL) | up to three years
  Quality of life will be assessed using the EORTC QLQ C30, EORTC QLQ Cr29 and Wexner score.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, Study Director — Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin J, Tang Y, Hu C, Jiang LM, Jiang J, Li N, Liu WY, Chen SL, Li S, Lu NN, Cai Y, Li YH, Zhu Y, Cheng GH, Zhang HY, Wang X, Zhu SY, Wang J, Li GF, Yang JL, Zhang K, Chi Y, Yang L, Zhou HT, Zhou AP, Zou SM, Fang H, Wang SL, Zhang HZ, Wang XS, Wei LC, Wang WL, Liu SX, Gao YH, Li YX. Multicenter, Randomized, Phase III Trial of Short-Term Radiotherapy Plus Chemotherapy Versus Long-Term Chemoradiotherapy in Locally Advanced Rectal Cancer (STELLAR). J Clin Oncol. 2022 May 20;40(15):1681-1692. doi: 10.1200/JCO.21.01667. Epub 2022 Mar 9. PMID 35263150